CLINICAL TRIAL: NCT02348229
Title: Effect of Enhanced Recovery After Surgery (ERAS) on C-reactive and Visceral Proteins in Patients With Advanced Gastric Cancer
Brief Title: Effect of Enhanced Recovery After Surgery (ERAS) on C-reactive and Visceral Proteins
Acronym: ERASAG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-212
Record Dates: First submitted 2015-01-17; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Gastric Cancer
Keywords: Enhanced recovery after surgery; laparoscopic gastrectomy; advanced gastric cancer; C-reactive,visceral proteins
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERAS group (Experimental): ERAS protocols
  Interventions: Procedure: ERAS protocols
- conventional pathway group (Other): using conventional pathway
  Interventions: Procedure: conventional pathway group

INTERVENTIONS:
Procedure: ERAS protocols — Normal meal allowed until 6 h before surgery and Carbohydrate drink until 2 h before surgery
  Arms: ERAS group
Procedure: ERAS protocols — No bowel preparation
  Arms: ERAS group
Procedure: ERAS protocols — No nasogastric placement; if used, remove on the 1st postoperative day
  Arms: ERAS group
Procedure: ERAS protocols — Vasoactive drugs used if need be
  Arms: ERAS group
Procedure: ERAS protocols — Temperature management
  Arms: ERAS group
Procedure: ERAS protocols — Intra-abdominal drains not to be used
  Arms: ERAS group
Procedure: ERAS protocols — Intraperitoneal Ropivicaine infusion
  Arms: ERAS group
Procedure: ERAS protocols — On the 1st postoperative day Nasogastric catheter removed /Urinary catheter removed.
  Oral non-opioid analgesia/Drinking 0.5L liquid. Active mobilisation
  Arms: ERAS group
Procedure: ERAS protocols — On the 2nd postoperative day：Drains removed Oral diet was initiated
  Arms: ERAS group
Procedure: ERAS protocols — 3-4th postoperative day： Stop oral non opioid analgesia
  Arms: ERAS group
Procedure: ERAS protocols — On the5-6th postoperative day Check discharge criteria
  Arms: ERAS group
Procedure: conventional pathway group — No solid foods at dinner before surgery and no liquids 12 h before surgery. Routine bowel preparation Nasogastric placement on the morning of surgery
  Arms: conventional pathway group
Procedure: conventional pathway group — Routine use of anesthesia medicine. Standard 5-trocar laparoscopy-assisted procedure. I.V. fluids not restricted (Ringer's lactate 20 ml/kg in the first hour, then at the rate of 10-12 ml/kg/h) Routine use of abdominal drainage tubes and placement of catheters.
  Arms: conventional pathway group
Procedure: conventional pathway group — 1st postoperative day: Keep Nasogastric catheter Removal of urinary catheter Opioid analgesic by intramuscular injection Parenteral nutrition until flatus. I.V. fluids not restricted Mobilization in bed
  Arms: conventional pathway group
Procedure: conventional pathway group — 2nd postoperative day Patient is advised to get out of bed until 24-48h after surgery
  Arms: conventional pathway group
Procedure: conventional pathway group — 3-4th postoperative day： Remove nasogastric tube after flatus Oral liquids started. Encouraged to walk in the ward.
  Arms: conventional pathway group
Procedure: conventional pathway group — 5-6th postoperative day：Oral diet was changed from liquids to semi-fluids and normal food.
  Drains removed
  Arms: conventional pathway group

SUMMARY:
The investigators designed a prospective randomized, controlled clinical trial then recruited 149 consecutive advanced gastric cancer patients. Further divided into a ERAS group (n=73) and a conventional pathway group (n=76). Surgical technique in both groups was same laparoscopic-assisted gastrectomy with D2 lymphadenectomy. Compared outcomes included clinical parameters and serum indicators.

DETAILED DESCRIPTION:
Enhanced recovery after surgery combined with laparoscopic-assisted gastrectomy was successfully carried out in this study. Recovery parameters such as the length of time to return to normal diet,mean hospital stay (d) were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Diagnosis confirmed by the endoscopic biopsy and total-body CT scan
3. No history of the chronic renal disease ,chronic liver disease, cardiopulmonary dysfunction, ASA score≦3
4. No neoadjuvant chemotherapy and radiotherapy
5. No digestive obstruction and distant metastasis

Exclusion Criteria:

1. Conversion to open gastrectomy
2. A large amount of bleeding leading(>500ml)
3. Patients withdrew their consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Compartition of postoperative hospital stay | up to 30 days after the operation

SECONDARY OUTCOMES:
Change from baseline in C-Reactive Protein( CRP) and visceral proteins level | baseline and 5 days
  1day before and 1-5days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, Doctor, Study Director — The First Hospital of Jilin University

REFERENCES:
- [Derived] Mingjie X, Luyao Z, Ze T, YinQuan Z, Quan W. Laparoscopic Radical Gastrectomy for Resectable Advanced Gastric Cancer Within Enhanced Recovery Programs: A Prospective Randomized Controlled Trial. J Laparoendosc Adv Surg Tech A. 2017 Sep;27(9):959-964. doi: 10.1089/lap.2016.0057. Epub 2016 Nov 22. PMID 27875094